CLINICAL TRIAL: NCT07143136
Title: Short-Term Outcomes of Early Administration of Colchicine in Non-ST Segment Elevation Myocardial Infarction Patients Treated With Drug-Eluting Stents.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, David Gamal William Ibrahim, Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ColchicineInNSTEMI2025
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Non ST-Segment Elevation Myocardial Infarction
Keywords: Colchicine; Inflammation; Non-STEMI
MeSH Terms: conditions — Inflammation; Non-ST Elevated Myocardial Infarction | interventions — Colchicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine group (Active Comparator)
  Interventions: Drug: Colchicine
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Administration of Colchicine 1 day before and 90 days after PCI in Non-STEMI Patients
  Arms: Colchicine group
Drug: Placebo — Matching Placebo Regimen
  Arms: Control group

SUMMARY:
Inflammation plays a central role in the pathophysiology of atherosclerosis and in the progression of coronary artery. Colchicine, an anti-inflammatory agent traditionally used for gout and pericarditis, has emerged as a potential therapy in cardiovascular disease due to its ability to inhibit microtubule polymerization and suppress interleukin-1β and the NLRP3 inflammasome pathway.

COLCOT and LoDoCo2 trails have demonstrated the efficacy of colchicine in reducing cardiovascular events in patients with coronary artery disease.

However, more recent trials, including OASIS 9 and COVERT-MI trials did not support the use of a short-term colchicine treatment at the acute phase of ST segment elevation myocardial infarction (STEMI) to reduce infarct size and improve outcomes. Limited data exist on the peri-procedural use of colchicine in non-ST elevation myocardial infarction patients undergoing PCI.

This study proposes to assess whether a loading dose of colchicine before PCI, followed by 3-months maintenance therapy, can improve short-term clinical outcomes and inflammatory markers in non- STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Non-STEMI
* Undergoing PCI with drug-eluting stents

Exclusion Criteria:

* Severe renal or hepatic dysfunction
* Colchicine hypersensitivity
* Active infection and active diarrhea.
* Gastrointestinal intolerance
* Pregnancy or breastfeeding.
* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE (composite of cardiovascular death, non-fatal MI, stroke, urgent revascularization) at 30 days and 6 months. | 6 months

SECONDARY OUTCOMES:
Rate of gastrointestinal side effects and other colchicine-related adverse events. | 3 months
Change in CRP from baseline to 3 months post-PCI | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Condello F, Sturla M, Reimers B, Liccardo G, Stefanini GG, Condorelli G, Ferrante G. Association Between Colchicine Treatment and Clinical Outcomes in Patients with Coronary Artery Disease: Systematic Review and Meta-analysis. Eur Cardiol. 2021 Oct 21;16:e39. doi: 10.15420/ecr.2021.31. eCollection 2021 Feb. PMID 34777579
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; ESC Scientific Document Group. Fourth universal definition of myocardial infarction (2018). Eur Heart J. 2019 Jan 14;40(3):237-269. doi: 10.1093/eurheartj/ehy462. No abstract available. PMID 30165617
- [Background] Mewton N, Roubille F, Bresson D, Prieur C, Bouleti C, Bochaton T, Ivanes F, Dubreuil O, Biere L, Hayek A, Derimay F, Akodad M, Alos B, Haider L, El Jonhy N, Daw R, De Bourguignon C, Dhelens C, Finet G, Bonnefoy-Cudraz E, Bidaux G, Boutitie F, Maucort-Boulch D, Croisille P, Rioufol G, Prunier F, Angoulvant D. Effect of Colchicine on Myocardial Injury in Acute Myocardial Infarction. Circulation. 2021 Sep 14;144(11):859-869. doi: 10.1161/CIRCULATIONAHA.121.056177. Epub 2021 Aug 23. PMID 34420373
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Martinez GJ, Celermajer DS, Patel S. The NLRP3 inflammasome and the emerging role of colchicine to inhibit atherosclerosis-associated inflammation. Atherosclerosis. 2018 Feb;269:262-271. doi: 10.1016/j.atherosclerosis.2017.12.027. Epub 2017 Dec 25. PMID 29352570
- [Background] Libby P. Inflammation in atherosclerosis. Arterioscler Thromb Vasc Biol. 2012 Sep;32(9):2045-51. doi: 10.1161/ATVBAHA.108.179705. PMID 22895665